CLINICAL TRIAL: NCT01729598
Title: Safety And Target Engagement Of Clu1 By Valproic Acid In Subjects With Intact Cognition: Proof Of Concept For The Development Of A Prevention Trial For Alzheimer's Disease
Brief Title: Valproic Acid in Subjects With Intact Cognition - Proof of Concept Study
Acronym: VPA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Gregory Jicha, 323-5550 (Other)
Collaborators: University of Kentucky (Other); Kentucky Alzheimer's Center (Unknown)
Responsible Party: Sponsor-Investigator, Gregory Jicha, 323-5550, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 12-0068-F6A
Record Dates: First submitted 2012-05-14; First posted 2012-11-20 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Alzheimer's Disease
Keywords: cognitively normal elderly population; safety and tolerability
MeSH Terms: conditions — Alzheimer Disease | interventions — Valproic Acid; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valproic Acid (Experimental): Valproic acid 250 mg or 500mg by mouth twice daily.
  Interventions: Drug: Valproic Acid
- Placebo (Placebo Comparator): Placebo capsule by mouth twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valproic Acid — generic valproic acid tablets packaged in placebo-matched capsules.
  Other Names: VPA; Depakote
  Arms: Valproic Acid
Drug: Placebo — Placebo capsule without active study medication in identical capsules as experimental medicine.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety of administration and effects of valproic acid on clusterin expression in cognitively-intact, healthy, elderly subjects. Clusterin mutations have recently been identified as a risk factor for the development of Alzheimer's Disease and changes in clusterin expression are seen in the elderly who develop Alzheimer's disease irrespective of whether they carry these genetic mutations or not. Valproic acid may prevent or reverse these changes.

Fourteen subjects with normal memory and thinking will participate in this study. Ten of these subjects will receive valproic acid and 4 will receive a "placebo" capsule with no active medicine. Participants will take study medication or placebo for 28 days and be followed for a total 35 days in this trial.

DETAILED DESCRIPTION:
This is a placebo-controlled, single-center, multiple ascending dose study. Seven healthy volunteers will be enrolled into 2 sequential cohorts, for a total of 14 enrolled subjects. The study will be conducted using two doses of valproate (250 mg PO bid, followed by 500 mg PO bid). At each dose level, 7 cognitively intact normal elderly subjects will be entered into the study with two subjects randomly selected to receive placebo while the other five subjects receive the designated dose of valproate.

Study procedures will include routine assessment of adverse events, safety labs, baseline MRI, physical and neurological exams, and cerebrospinal fluid collection.

Other investigational medication or devices are prohibited during this study.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged 65-90, inclusive.
2. English-speaking, to ensure compliance with cognitive testing and study visit procedures.
3. Female participants must not be pregnant or of childbearing potential, i.e. either surgically sterile or postmenopausal for > 1 year.
4. Stable medical condition for three months prior to screening visit, with no clinically significant abnormalities of hepatic, renal, and hematologic function defined as follows:

   * Platelets > 100,000
   * Serum creatinine ≤ 1.6 mg/dL
   * Liver function tests ≤ 1.5 upper limit of normal
   * No clinically significant abnormalities of other laboratory studies (blood counts, chemistry panel, urinalysis) as determined by the study physician
5. Stable medications for 4 weeks prior to screening visit.
6. Able to ingest oral medications.
7. No history of adverse drug reactions to VPA or similar agents.
8. Physically acceptable for this study as confirmed by medical history, physical exam, neurological exam and clinical tests in the opinion of the study physician.
9. Not demented by Hachinski Ischemic Index (< 4).

Exclusion Criteria:

1. Significant neurologic disease such as Parkinson's disease, stroke, brain tumor, multiple sclerosis or seizure disorder.
2. Major depression in past 12 months (DSM-IV criteria), major mental illness such as schizophrenia, or recent (in past 12 months) alcohol or substance abuse by history.
3. History of invasive cancer within the past two years (excluding non-melanoma skin cancer).
4. Contra-indications to lumbar puncture (bleeding disorder, platelet count < 100,000, anticoagulant treatment, major structural abnormality or sepsis in the area of the lumbosacral spine that would make spinal fluid collection technically difficult).
5. Clinically significant MRI abnormalities that contraindicate lumber or suggest central nervous system disease processes that could influence study outcomes in the opinion of the PI.
6. Use of any investigational agents within 30 days prior to screening.
7. Major surgery within eight weeks prior to the Baseline Visit.
8. Severe unstable medical illnesses, including uncontrolled cardiac conditions or heart failure (New York Heart Association Class III or IV) .
9. Antiretroviral therapy for human immunodeficiency virus (HIV).
10. Residence in a skilled nursing facility.
11. Blindness, deafness, language difficulties or any other disability which may prevent the participant from participating or cooperating in the protocol.

Excluded Medications

1. Experimental drugs
2. Lamictal
3. Tricyclic antidepressants (amitriptyline/nortryptiline)
4. Carbamazepine/ oxcarbazepine
5. Benzodiazepines
6. Phenobarbital
7. Phenytoin
8. Tolbutamide
9. Topiramate
10. Warfarin
11. Zidovudine

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Estus, PhD, Principal Investigator — University of Kentucky; Gregory Jicha, MD, Principal Investigator — University of Kentucky
Locations (1):
- Sander's Brown Center on Aging, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with interested investigators that submit a data request to the UK Alzheimer Center Biostatistics Group upon publication of the primary manuscript from this study. The request will be reviewed for scientific validity and human subjects protection issues prior to approval for release. IPD that may be released includes all clinical data stripped of identifying information. Clinical Information will be assigned a blinded subject number that protects the identity and HIPAA protected information collected as part of this study. To request data, follow the instructions at the following link: http://www.uky.edu/coa/adc/investigators-research-resources
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1/1/19 to 12/31/28
Access Criteria: Access will be granted to any investigator upon provision of an acceptable project hypothesis and specification of data desired. Oversight by the project team will ensure that redundant projects do not result in competitive use of the resources. Project data access will be determined by the PI and investigator team at UK within these broad access terms. There will be no cost for data access. We stipulate that the parent grant UL1TR001998 should be cited by those with whom data is shared.
URL: http://www.uky.edu/coa/adc/investigators-research-resources

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valproic Acid | Placebo
Started | 10 | 4
Completed | 10 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valproic Acid | Placebo | Total
Number analyzed (Participants) | 10 | 4 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 10 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (7.3) | 81 (12.2) | 78 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 6 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 4 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 4 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events Over the Duration of the Study by Study Arm
Description: Safety assessments will be based on medical review of adverse event reports and the results of vital sign measurements, physical examinations, and clinical laboratory tests throughout the study. The incidence of observed toxicities and adverse events will be tabulated, the frequencies compared in participants who receive active medication and those who receive placebo, and reviewed for potential significance and clinical importance.
Time Frame: Day 35
Measure: Count of Participants; unit: Participants
Arm/Group | Valproic Acid | Placebo
Number analyzed (Participants) | 10 | 4
Participants | 8 | 1

2. Primary Outcome: Change in Cerebrospinal Fluid Amyloid Levels (pg/ml) Over 28 Day Intervention Period by Study Arm
Description: Change in cerebrospinal fluid amyloid-beta 1-42 levels in pg/ml from baseline to end of treatment (day 28)
Time Frame: Baseline and day 28
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Valproic Acid | Placebo
Number analyzed (Participants) | 10 | 4
pg/ml | 57.1 (28.4) | 44.7 (24.9)
Statistical Analysis 1: Comparison: Valproic Acid vs Placebo; Test type: Superiority; p = 0.55, t-test, 2 sided

3. Secondary Outcome: Change in Cerebrospinal Fluid P-tau Levels (pg/ml)
Description: Change in cerebrospinal fluid p181-tau levels (pg/ml) from baseline to end of treatment (Day 28)
Time Frame: Baseline and day 28
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Valproic Acid | Placebo
Number analyzed (Participants) | 10 | 4
pg/ml | -5.7 (11.9) | 11.0 (25.7)
Statistical Analysis 1: Comparison: Valproic Acid vs Placebo; Test type: Superiority; p = 0.19, t-test, 2 sided

4. Secondary Outcome: Change in Free & Cued Selective Reminding Test- Free Recall (Number of Items Correct)
Description: Change in Free & Cued Selective Reminding Test- delayed free recall from baseline to end of treatment (Day 28)
Time Frame: Baseline and day 28
Measure: Mean (Standard Deviation); unit: number of items recalled
Arm/Group | Valproic Acid | Placebo
Number analyzed (Participants) | 10 | 4
number of items recalled | 1.4 (3.5) | -4.5 (3.4)
Statistical Analysis 1: Comparison: Valproic Acid vs Placebo; Test type: Superiority; p = 0.02, t-test, 2 sided

5. Secondary Outcome: Change in Cerebrospinal Fluid Clusterin Levels (pg/ml)
Description: Change in cerebrospinal fluid clusterin levels (pg/ml) from baseline to end of treatment (Day 28)
Time Frame: Baseline and day 28
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Valproic Acid | Placebo
Number analyzed (Participants) | 10 | 4
pg/ml | 2610 (4373) | 201 (871)
Statistical Analysis 1: Comparison: Valproic Acid vs Placebo; Test type: Superiority; p = 0.31, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 35 days
Arm/Group | Valproic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/4
Other Adverse Events (participants affected / at risk) | 8/10 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valproic Acid (N=10) | Placebo (N=4)
hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0)
fatigue (Nervous system disorders) | 3 (4) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No